CLINICAL TRIAL: NCT03816046
Title: The Quadrant vs the Six Injection Technique in Primary Focal Hyperhidrosis Using Botulinum Toxin: a Cross-over Clinical Trial.
Brief Title: Hyperhydrosis Treatment Using Botulinum Toxin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St Joseph University, Beirut, Lebanon (Other)
Responsible Party: Principal Investigator, samer jabbour, M.D, St Joseph University, Beirut, Lebanon
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: usj-05
Record Dates: First submitted 2017-06-12; First posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Hyperhidrosis
Keywords: botulinum toxim; abobotulinum; hyperhydrosis; injection
MeSH Terms: conditions — Hyperhidrosis | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: describe two safe and reproducible techniques for the treatment of hyperhidrosis using botulinum toxin. The same patient will receive two different injection technique in each armpit and will be evaluated subjectively and objectively.
Who Masked: Outcomes Assessor
Masking Description: the objective assessment with iodine starch test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Technique 1 The Quadrant technique (Experimental): Intervention: 25 Botulinum Toxin injections. 5 vertical lines and 5 horizontal lines will be draw on the hair bearing area of the armpit amounting to 25 injection points being more concentrated on the center. Each injection consists of 5Units of abobotulinum
  Interventions: Drug: botulinum toxin A
- Technique 2 the six injection technique (Experimental): Intervention: 6 Botulinum Toxin injections. will consist on 6 injections in the hair bearing area equally spaced with each consisting of 8units
  Interventions: Drug: botulinum toxin A

INTERVENTIONS:
Drug: botulinum toxin A — injection in hair bearing area of armpits

SUMMARY:
The purpose of this study is to describe two safe and reproducible techniques for the treatment of hyperhidrosis using botulinum toxin. The same patient will receive two different injection technique in each armpit and will be evaluated subjectively and objectively.

DETAILED DESCRIPTION:
The abobotulinumtoxinA (ABO) will be used in all patients. The ABO will be prepared by adding 4 cc of normal saline to a 500-unit Dysport© (Ipsen Ltd, Berks, UK) vial Preinjection patient pictures will be taken showing the technique used for each armpit.

Injection technique:

1. Technique 1 The Quadrant technique: 5 vertical lines and 5 horizontal lines will be draw on the hair bearing area of the armpit amounting to 25 injection points being more concentrated on the center. Each injection consists of 5Units of abobotulinum
2. Technique 2 the six injection technique: will consist on 6 injections in the hair bearing area equally spaced with each consisting of 8units

Follow up will be done at 15 days for post injection pictures with iodine starch test A total of 15 male patients will be recruited. And the injection for each armpit in a given patient is randomized.

ELIGIBILITY:
Inclusion Criteria:

Consecutive 15 male patients presenting to our clinic for primary localized hyperhidrosis will be included in this study

Exclusion Criteria:

* Patient that has received a botulinum injection in the past year

Patient that had a liposuction in the armpit or laser for the hair

Patients with preexisting neuromuscular conditions (myasthenia gravis, Eaton Lambert syndrome) Patients using medication that could potentiate the effect of botulinum (ex: aminoglycoside antibiotics) Patients with sensitivity to botulinum toxin or human albumin

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
objective iodine startch | 3weeks
  Objective assessment will be done using the iodine starch after a 5 min jumping jack on the post injection visit.

SECONDARY OUTCOMES:
subjective: patient satisfaction | 3 weeks
  Patient satisfaction will be determined by a questionnaire completed at 3 weeks post-treatment. Subjects will indicate how satisfied they are on a 4-point scale (1-4) as follow:
  1. Very Satisfied
  2. Satisfied
  3. Dissatisfied
  4. Very Dissatisfied.
subjective: pain on injection | day 0
  A verbal scale from 1-10 will be addressed for every patient and every armpit

CONTACTS AND LOCATIONS:
Locations (1):
- Hotel Dieu de France, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No